CLINICAL TRIAL: NCT02341690
Title: The Effectiveness of Smartphone Delivered Interval Walking Training on Physical Activity and Glycemic Control in Patients With Type 2 Diabetes: a Pragmatic Randomized Controlled Trial - Part of The InterWalk Study
Brief Title: Intervention Study - Effectiveness of Smartphone Delivered Interval Walking Training to Patients With Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: Center for Physical Activity Research (CFAS) (Unknown); The Danish Center for Strategic Research on Type 2 Diabetes (Other); The Danish Diabetes Association (Other); The Parker Institute, Department of Rheumatology, Copenhagen University Hospital at Bispebjerg and Frederiksberg. (Unknown)
Responsible Party: Principal Investigator, Laura Staun Valentiner, PhD-student, University of Copenhagen
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: INTERWALK
Record Dates: First submitted 2015-01-09; First posted 2015-01-19 (Estimated); Last update posted 2018-05-24 (Actual); Status verified 2018-05

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Type 2 diabetes; Interval Walking Training; Motivation
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Active Comparator): Standard rehabilitation with exercise
  Interventions: Other: control
- Intervention (Interval Walking Training) (Experimental): Interval Walking Training with the InterWalk app, 3 times per week, 60 min. per sessions for 52 weeks. The intervention period is divided into
  1. a period that follows standard care in the municipality (from 8-14 weeks according to the municipality.
  2. a period (from week 8-14 to week 52) the patients will do Interval Walking on their own.
  3. After the intervention at the promotion centre (8-14 weeks), the intervention group will be divided into to groups - a Interval Walking group (IWT) and a Interval Walking group with support (IWTsupport).
  IWTsupport: Patients in this group (after intervention at the promotion centre) will in addition to the IWT receive motivational support from week 8-14 to week 52 by the health professionals at the promotion centre.
  Interventions: Other: Interval walking training

INTERVENTIONS:
Other: Interval walking training — Interval Walking Training with the InterWalk Application An Interval-walking bout will consist of repeated cycles of 3 minutes of fast and 3 minutes of slow walking at 70% and 40% of the smart-phone assessed peak VO2-rate, respectively.
  IWT is conducted for at least 60 minutes per day, three days per week. Compliance is monitored continuously using the on-board accelerometer logger
  Arms: Intervention (Interval Walking Training)
Other: control — Standard care at the promotion centre in the municipality
  Arms: Control

SUMMARY:
Type 2 Diabetes (T2D) is one of the most common chronic diseases world vide. Patients with T2D experiences reduced quality of life and have a lower physical activity level. Physical activity is well documented treatment to the patient group. The effect of physical activity is shown to reduce co-morbidity, and better functional level and quality of life.

Interval Walking Training (IWT) is a new and effective exercise type. IWT is done by walking in a slow and a fast tempo. InterWalk is an application to a smartphone. By using InterWalk the patient can to IWT independently and when used, the app has, as an exercise tool, the potential to better the individual functional level and to measure the physical activity level with the integrated personalised walking test.

Motivation for change of habits and lifestyle is subjectively determined by the individual, his or hers individual resources and environment. It is important to get insight in these individual challenges in order to be better structure possible help.

The combination of an exercise log, a measure of physical activity fromInterWalk and insight in motivational aspects on an individual level, is essential for successful individualised training.

The primary objective of the study is to investigate if the InterWalk app is more effective in increasing the physical activity level compared to a standard care offer in a sample of newly T2D diabetes patients across 52 weeks.

Secondarily, we will investigate if the IW app can reduce sitting time, induce weight loss, improve glycaemic control, increase quality of life, improve cardio-respiratory fitness and reduce the use of diabetes medication.

The study is designed to test the hypothesis that replacing a standard exercise program in the normal municipal standard care with the Interval Walking Training delivered by the IW app with and without a motivational support program, can increase the long-term physical activity level in patients with T2D for a period of 52 weeks.

From January 2015 to June 2016 all patient's with T2D, who are referred to the promotion centres in the municipality, will be offered to participate in the study. In total 513 patients with T2D from different municipalities in Denmark will be included and randomly allocated into three groups. One group will receive standard care and the two other groups will do IWT with the InterWalk app. All three groups are followed by the promotion centre for 8-14 weeks (according to the rehabilitation in the municipality) and hereafter only one of the IWT groups will receive motivational support up to 52 weeks.

All patients, no mater group allocation, will be tested and fulfill questionnaires, three times during the intervention period - at baseline, after 8-14 weeks and after 52 weeks. The interventions take place at the promotion centres in the municipalities two times a week and the patient will be encouraged train by them selves one time a week.

DETAILED DESCRIPTION:
Background Type 2 diabetes (T2D) is one of the most common long-term medical conditions worldwide. The patients have a two-fold increased mortality rate compared to the general population T2D is a major problem in Denmark and the incidence is estimated to rise from 280.000 today to approximately 500.000 people by 2020 (5).

The T2D rehabilitation program in the Danish municipalities has the overall purpose of introducing and helping patients to a healthier lifestyle (6). The program is conducted in a period of 8-14 week with some or no exercise intervention, with no long-term follow-up. Not much is known on the amount and integration of PA in the patient's everyday life following the intervention (7). This major variation across municipalities poses a problem in the rehabilitation of TD2, as the quality of rehabilitation depends on the geographical location of the T2D patient.

Several studies have shown that supervised PA is advantageous; in patients with T2D on key metabolic factors (6-9) and that it improves quality of life and reduces the risk of all-cause mortality (1,2,6,10,11,12). Due to the many beneficial effects of PA on T2D patients, PA is an important factor in the prevention and treatment of T2D (13). Long-term PA interventions have employed supervised exercise regimes (14,15) that are effective, but also demanding and expensive. Attempts to increase the daily physical activity level on a large scale, in a free-living "real life", have very little effect (14-16) despite well-established patient education programs. In general, the exercise adherence is low and dropout rates are high in this group of patients. A large number of patients with T2D experience diminished quality of life, decreased physical functioning, diminished exercise tolerance (17), numerous patients are unmotivated or incapable to change behaviour and the prevalence of depressive and anxiety symptoms are highly prevalent in T2D patients (17,18,19). Collectively this could pose important barriers to engagement in exercise and reaching the recommended level of PA (20).

Karstoft et al (2013) examined the feasibility of implementing a free-living interval walking (IWT) and continuous walking training program in a smaller sample of patients with T2D. IWT was initiated and monitored by a Japanese training device, the JD-mate (10). The study found remarkable effects on physical fitness level, body composition and glycaemic control and with a compliance rate of more than 85% and a very low dropout level (9). Based on the experiences by Karstoft et al and several pilot testing's in the Danish Diabetes Association (DF), we believe that IWT can be an approach to handle lack of PA in patients with T2D. However the JD-mate, is expensive (3500 kr.), Japanese instructions, lacks automatic transmission of data and is thus not user-friendly on a larger scale. It is evident that novel low cost, more sustainable exercise solutions and suitable vehicle are needed and through this, improve quality of life and increase life expectancy in these patients.

The use of Tele-Health interventions (THI) have the potential to educate and engage patients with T2D in self-management in the long-term and the evidence suggests that THI could be effective and feasible in improving clinical outcomes in diabetes care (14,15,22,23). The widespread and increasing use of smartphone applications is opening new ways to improve health and health care delivery. It might be ideal to use THI to increase physical activity and hereby target a large part of the population by simple and inexpensive means. The smartphone has been used as a tool among others to register exercise, diet, weight and plasma glucose levels, but the evidence of using a smartphone as an exercise device is lacking (24).

In 2010 the Danish Centre for Strategic Research in Type 2 Diabetes (DD2) and TrygFondens Centre for Aktiv Sundhed (CFAS), Rigshospitalet, Denmark, developed the InterWalk Application (IW app) to the smartphone to promote IWT on a larger scale. IWT has the potential to increase physical activity in a large group of T2D patients and hopefully improve lifestyle in patients with T2D. However, motivation for lifestyle changes is subjectively driven and individually determined (25-27). The personal resources and the close environment are key determinants of how challenges are handled in everyday life (28,29). Motivational factors are important for changing physical activity behaviour in patients with T2D, but knowledge on how motivation is maintained for a sustainable active lifestyle is limited. Studies of the effectiveness of employing smartphones as a vehicle to improve physical activity behaviour in everyday life in the long-term in patients with T2D is therefore needed.

Aim/purpose - (Hypothesis) The primary objective of the study is to investigate if the InterWalk app is more effective in increasing the moderate-and-vigorous physical activity level compared to a standard care offer in a sample of T2D patients across 52 weeks.

Secondarily, we will investigate to what extend the IW app can reduce sitting time, induce weight loss, improve glycaemic control, increase quality of life, improve cardio-respiratory fitness and reduce the use of diabetes medication.

The primary hypothesis is to test the hypothesis, that replacing a standard exercise program in the normal municipal standard care with the Interval Walking Training delivered by the IW app, the patient will become more physical active. The secondary and explorative hypothesis is that motivational support will increase the individual long-term physical activity level in everyday in patients with T2D.

Methods Study design The study is a 52-weeks single-blinded pragmatic randomized controlled trial, where the participants are allocated into three arms. Two of the arms will receive IWT with or without additional support. The control arm will receive the standard care. The interventions are delivered by the Danish municipalities. A detailed description of the three arms is found below. The study is carried out in a subgroup of the DD2 cohort.

Participants, Recruitment and eligibility All patients referred to the promotion centre in the municipalities from January 2015 will be screened for eligibility. The patients will be informed about the study and will be given formalized oral and written material, a consent form and a free post envelope. Upon reception of the consent form by the health professional at the municipality, the patient will be contacted by one of the health professionals assigned to the study and a date for the first visit is arranged.

Enrolment is anticipated to take approximately 18 month and begins in January 2015, and is expected to be completed in July 2017. The intervention will take place at the promotion centres in municipalities in Denmark.

Sample size considerations The minimum difference of interest (MDI) is 10 minutes per day. After applying Bonferroni adjustment due to multiple comparisons in the three group trial and shared end-points, a total of 393 participants are needed using an sample SD of 25 minutes per day (30) with an α of 0.017 (two-tailed) to obtain a statistical power (1-β) of 80%. Allowing for an attrition rate of 30%, 513 patients (171 in each group) are allocated in the three arms.

Allocation, randomization and concealment Patients are randomized using random permuted blocks (2x2x2) and stratified by gender to ensure an equal number of participants in all groups across the allocation period. The allocation sequence is generated through a standardized computer program by an independent researcher not affiliated to the study and is concealed until the study arms are assigned. Randomization of each patient to one of the three groups in the study is done after the baseline tests have been conducted by the health professionals at the promotion centres. The scientific staff is blinded to the allocation. The health professionals at the promotion centre are not blinded to allocation according to control group (1/3) or intervention groups (1/3: IWT and 1/3: IWTsupport). After the intervention period at the promotion centre, the allocation to either control, IWT or IWTsupport is unsealed to the patients and the health professionals at the promotion centres. The scientific staff is still blinded.

Interventions Group 1 (control group): Patients in this group will receive the standard rehabilitation program with the overall purpose of lifestyle changing in T2D patients in a multimodal setting in the municipality including physical activity. In addition to exercise, the rehabilitation consists of education, smoking cessation and dietary change with the purpose of weight loss, motivation groups and self-care. The duration of the rehabilitation differs between municipalities with duration from 8 to 14 weeks. There will be no follow-up from the municipality, which is the normal procedure in the municipality.

Group 2 (IWT with without motivational support after 8-14 weeks): Patients in this group will be engaged to IWT with the IW app (see: The InterWalk Application). The intervention period will follow the period in which the rehabilitation program is carried out in the municipality (duration from 8-14 weeks). The patients are encouraged to perform IWT three times per week, 60 minutes per session. The municipality offers to walk with the patient´s two times per week for 60 minutes per session in group sessions with additional 30 minutes of group discussion afterwards. The last and third time the patients have to walk by themselves for 60 minutes per session. The participating patients will receive a thorough introduction to the IW app and follow-up during the intervention (8-14 weeks) from the health professionals. At the end of the intervention period, the health professionals, conducts a transition program, preparing the patients to continue IWT with IW app on their own. There will be no follow-up from the municipality, which is the normal procedure in the municipality.

Group 3 (IWTsuppport) IWT with motivational support after 8-14 weeks: Patients in this group will like patient´s in intervention group 2 be engaged to IWT with the IW app. The intervention period will be 52 weeks. The first 8-14 weeks will be conducted together with group 2 with a thorough introduction to the IW app and IWT three times per week for 60 minutes. In addition to the IWT from week 0 to 52, the patients in this group will receive motivational support from week 8-14 to week 52 by the health professionals at the promotion centre (see below for information regarding the IW app and the motivational support part).

The InterWalk Application The IW App is a personal trainer as well as a monitor unit, which allows continuous and automatic transmission of physical activity data to a central data base in DD2. The IW app guides the user in IWT with repeated cycles of 3 minutes fast and slow walking. During IWT the app provides the patients with continuous feedback on the walking intensity (10). The feedback is personalized through a standardized eight-minute walking test, performed before engaging in IWT. The patients are able to track exercise history and receive historic feedback on the quality of the IWT sessions. The feedback system employs the on-board accelerometer and GPS system to assess intensity and geographical location.

The patients are obligated to enter their social security (CPR) number before using the app. Uniquely, this will allow the scientific teams to integrate the app into the health care system, link the data with the Danish disease and demographic registers and thus, will enable the study of long term nation-wide effects of IWT in T2D rehabilitation.

The application has been through extensive piloting in different groups of patients with T2D. Information on training intensity, total number of steps per day and IWT-data and data from the standardized walking test is stored on the smartphone or IPod and automatically transmitted to a central database when connected to Wi-Fi or mobile data network.

Individual motivation (IWTsupport) Motivational support will in addition to the IWT be offered in intervention group 2 after the intervention at the promotion centre. The support is initiated and conducted by the health professionals at the promotion centres.

* SMS-track: The patient i intervention group 2 will receive motivational support which consists of Short Message Service -Track (SMS-Track), phone calls, goal setting and i motivational interviews (see below). The different parts of the motivation intervention will be handled and executed by the health professionals at the promotion centres in the municipalities.
* Short Message Service - Track: The first Sunday after enrolment a SMS-track is send to all patients in either group 2 or 3. The patients will be asked to confirm that they are part of the study, before the next SMS regarding their IWT is send. The patient can receive up to 3 SMS's regarding IWT depending on their answers.
* Phone calls: The patient's answers to the SMS-track, constitute whether a personal phone call from a health professional if necessary. The aim of the call is to help and support the patient in continuing to keep doing IWT with IW app. Questions from the health professionals addresses how the patient is doing in general, why the patient has answered that they haven't been doing IWT the past week, questions regarding how to help the patient doing IWT, or questions about the IW app. The patient will have time to ask questions of concern to the health professional.
* Standardized walking test: Every 4th week a SMS will be send to the patient regarding new goal setting.

Individual goal setting: To measure the patients motivation for physical activity using the IW app in group 2 and 3, we ask the patients to set individual goals every 4th week, related to their everyday life, during the intervention period (group 2 (4-18 weeks) and group 3 (0-52 weeks) (40) - The goal setting is based on the S.M.A.R.T.-principle where S stands for Specific, M for Measurable, A for achievable , R for relevant and T for timely (41).

- IWTsupport group sessions: Patients in group 3 have the opportunity to participate in IWT with other patient and a InterWalk ambassador at the municipality once a week after the intervention at the promotion centre.

Motivational interviews: Four motivational interviews will be scheduled for patients in group 2, in the period where the patient no longer is part of the formalised IWT in the municipality (week 12-52). The aim of these interviews is to help he patients to maintain motivation and focus tin prioritizing IWT in their everyday life. The interview will take place at the promotion centre.

Measurements

* Level of daily physical activity To evaluate the level of moderate-to-vigorous-intensity physical activity all participants will be equipped with an accelerometer (Axivity AX3, Newcastle, UK) for 10 consecutive days, 3 times during the intervention period - at baseline and after 4-18 weeks and 52 weeks after enrolment. One accelerometer will be placed with patch (Leukomed T, BSN medical, Germany) on the lateral side of the right thigh and one accelerometer on the lumbar spine. The patients will be instructed not to remove the accelerometer during the three periods. The accelerometers can be worn when taking a shower, swimming etc.
* Smart-phone administered standardized walking test The walking test in the IW app consists of 5 stages; 1) 30 sec. of standing still, 2) 2 min. of slow walking 3) 2 min. of walking at moderate intensity 4) 2 min. walking at high intensity 5) 1 min. walking at highest intensity possible. The four later paces are self-selected. The test is performed with the Smartphone placed at a pocked at the hip and the instructions are communicated auditory through earphones. To ensure the right walking intensity in the intervention period, the patients are asked to perform the test every 4th week.
* Sit-to-Stand Test The test measures the lower body strength and will be administrated using a chair without arms, with a seat height of 43 cm. The patient is encouraged to complete as many full stands as possible within a 30-sec time limit (32).

Electronic log of data from IWT to the central database Adherence to the intervention is determined by an evaluation of the electronic log of data from IW app to a central database. All the uploaded data can be quantified into adherence.

* Physical Activity Questionnaire "The Resent Physical Activity Questionnaire" (RPAQ) is a self-rated physical activity questionnaire. The RPAQ has 9 main questions which covers 4 domains of physical activity: domestic life, work, recreation and transport. Physical Activity is estimated in MET (Metabolic Equivalent) (35).
* Short Form -12 (SF-12) The SF-12 was developed as a short form of the 36-item Short-Form Health Survey (SF-36). The questionnaire consists of 12 questions and uses a Likert scale of 1 to 3 for the physical function items; 1 to 5 for the bodily pain, social function, and general health perceptions items; 1 to 6 for the vitality and mental health; and a dichotomous scale of yes/no for the presence of role function limitations. The higher score, the higher level of health or functioning (34).
* Behavioural exercise regulation questionnaire (BREQ-2) Behavioural exercise regulation questionnaire (BREQ-2) measures individual motivation for physical activity. The Questionnaire consists of 19 questions in a 0-4 Likert format.
* Questions on motivation for physical activity for patients with Type 2 Diabetes All patients will be asked to answer four questions in a 0-4 Likert format, regarding their habits for doing physical activity after being diagnosed with T2D.
* Personality Questionnaires The patient will be asked to complete two questionnaire regarding personality, the NEO-Five Factor Inventory (NEO-FFI) and a Sensation Seeking Scale (SES).

The NEO-FFI consists of 60 questions in a 0-4 Likert format constructed by selecting 2 items from each of the six facets characterizing each of the five personality traits (Neuroticism, Extraversion, Openness, Agreeableness, Conscientiousness) assessed by NEO-PI-R (36).

The Sensation Seeking Scale is a 40 items self-administered questionnaire and consists of 40 questions designed to test the tendency towards varied, novel and intense sensations (37). The SES-questionnaire is in its design impertinent as it consists of only two possible response options for each question. The patient will be encouraged to answer the questions, but is not required an answer.

We do not know much about what characterizes the individual to either participate or to decline an intervention e.g. diet, smoking cessation or physical activity. The two personality questionnaires are part of the project because it is essential to get more knowledge on personality traits, risk behavior and adherence to an intervention in this case physical activity. By this knowledge it will be possible to better individualize the intervention and by this hopefully get a higher adherence in the long term.

* Monitoring of body temperature To detect possible effects of exercise on mitochondrial function a measure of body temperature with an ear thermometer will be performed. Time of measure, season and weather conditions, diseases within the last week and meals before the measure will be noted.
* Demographic and social economic Information: Information on demographic will be obtained using standard procedures (height, weight, waist and hip circumference). The demographic data will be obtained from the patient's journal at the Promotion Centre. A tape measure and a weight will be provided to each promotion centre to ensure standardization among health professionals.
* Relevant national registers will be used for information regarding co-morbidities, medical history and use of medicine. All the information from the patient's journal and from relevant registers will be used when all data, from all patients, are collected. The data will be protected by the "Lov om behandling af personlige oplysninger" (see 'Protection of personal information', page 12).
* Metabolic markers The patients are encouraged to maintain the recommended regular visits every 3th month at the general practitioner (GP) in the intervention period (52 weeks). Results from the visits including the blood sample are collected from the national database DSAM.

Risk, side effects, and discomfort General considerations The exercise intervention (Interval Walking Training) is expected as a minimum to be as effective as the standard care programme currently offered to patients with T2D at the municipality. Interval walking Training with the use of a Tele-Health solution is providing patients with T2D with a feasible option on how to implement and maintain a physical active lifestyle in a gentle and flexible way. The intervention is expected to result in remarkably health benefits on a long-term basis in terms of improved increased VO2max, blood glucose regulation, and quality of life and motivation for a more active everyday life.

The study is important and will contribute to great knowledge about how to implement and thus increase public health in a large and growing cohort of patient´s with T2D.

Measurements Smartphone administered walking test: The patients are expected to reach 80-85% of VO2max during the IW walking test. This will cause some degree of breathlessness.

AX3 Axivity accelerometers: Due to the patched by which the accelerometers are hold on the thigh and lower bag, itching and redness may occur in allergic subjects. In those cases the subjects are encouraged to remove the patches immediately and if necessary consult a general practitioner. The patients will be informed on procedures in writing containing pictures of the application of accelerometers and possible discomfort.

Interval walking training: The IWT will cause some degree of breathlessness in the fast walking interval periods.

Anthropometric measurements, sit-to-stand test, temperature, questionnaires and motivational initiatives: These methods are not associated with any known risk or other unpleasant.

Statistical analysis All analyses will be conducted according to the Intention-to-treat principle. Mixed model analyses will be employed to determine the group X treatment effects of the intervention across twelve months. The secondary outcomes will be analyzed using the same approach. Assuming that the data on potential drop-outs are missing at random multiple imputation procedures will employed to handle missing data. Patterns of missing data will be investigated. Per protocol analyses will be performed to support the primary analysis.

Ethical considerations The study is expected to result in limited risks, adverse effects and discomfort to the patients. No invasive methods will be used besides blood samples taken by the GP at regular visits. The patients will benefit from the study in terms of enhanced physical capacity and by introduction to effective training methods.

The randomization of the participating patients into three groups is necessary to evaluate the effectiveness of the InterWalk app. The intervention groups (group 2 and 3) are alike as long as the standard rehabilitation with physical activity proceeds in the municipality. From hereafter only group 3 will be supervised and will receive motivational support from the health professionals. This differentiation between groups is needed in order to obtain insight regarding motivational factors of importance to the individual, to maintain a physical active everyday life.

The two personality questionnaires in the study will help to get insight on personality, physical activity and motivation for behavioural changes (e.g. more physical active everyday life). With this knowledge, the results from the study can help the health professionals at the promotion centres, to better allocate patients with T2D, into a rehabilitation offer adjusted to the individual and not as a standard offer in the municipality.

Expected outcomes Performing IWT might be a suitable and effective way to exercise for at large group of patients with T2D. The patient can walk everywhere and IWT can hereby be integrated and maintained in the patient's everyday life. Experiences from the study can be used in planning interventions with the IW app and IWT, to patients with other lifestyle diseases e.g. Constructive Obstructive Pulmonary Lung Disease (COPD) and Heart Diseases. The aim is to obtain lifelong physical activity for the individual in their everyday life.

Patient insurance The intervention takes place at the promotion centres in the Municipality and the patient is, if anything should happen during the intervention period, insured by 'Patient Forsikringen'. The law says '…personer, der deltager i biomedicinske forsøg m.v., der udføres af private firmaer, foreninger m.v. er omfattet af lovens område, hvis forsøget udføres under direkte ansvar af et sygehus, en statslig højere uddannelsesinstitution m.fl.'. The University of Copenhagen is the 'statslige højere uddannelsesinstitution in this study.

Protection of personal information All personal information on the patient's identities are protected by the "Lov om behandling af personlige oplysninger". A unique subject ID number will be subscribed to all patients in order to anonymize data. The identification key (ID to personal information) will be encrypted and stored securely and separately from the unique ID number on a secure database. In this way no information on patient´s can be assigned to the ID number. All data is automatically backed up on a secure server. Questionnaires is completed online and automatically uploaded with the ID number to the secure data base.

Each promotion centre will be assigned with secured logons to the database and only the health professional assigned to the study, will get logons and will only be able to see the patients included in the study at their promotional centre. The scientific members have access to the secure database and data from all the included patients. All data will be secured in the database and a bag up of all the data is stored in an extern hard disk which is also secured. It is possible to track all logons to the database as well as all tasks done in the database.

To enter the IW app the patients are obligated to enter their CPR number, which immediately are encrypted to protect against inappropriate use of the number from unauthorised people not connected to the study. The health professionals in the municipalities will be educated in data entry and will only have access to their own promotion centre. Only the research team will have access to data processing.

The IW app is already approved by "Datatilsynet" (2008-58-0035 (paraplygodkendelse i Region Syddanmark)) and the RCT-study will in addition be reported to "Datatilsynet".

Compensation There will be no compensation given to the patient. All participating patients are treated in accordance with the national guidelines regarding rehabilitation in the municipality.

Dissemination The data will be published in international peer-reviewed journals. The results are to be reported according to the CONSORT guidelines (38). All results will be disseminated (negative, positive and inconclusive findings). All result will be published (positive, negative and inconclusive).

For references - see the section 'References'

ELIGIBILITY:
Inclusion Criteria:

* Patients are eligible if they are diagnosed with T2D and are more than 18 years of age.

Exclusion Criteria:

* Medical contraindications to exercise e.g. if the patient has developed chronic complications in the locomotive apparatus, e.g. painful osteoarthritis or heart conditions (30,39) and already is participating in other studies at the promotion centres concerning PA.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 226 (Actual)
Dates: Start 2015-01; Primary Completion 2017-12-17 (Actual); Study Completion 2017-12-17 (Actual)

PRIMARY OUTCOMES:
Changes in Physical activity from baseline to 52 weeks, measured with accelerometrics | 52 weeks
  Physical activity is measured with accelerometrics, where the patient wear two accelerometers (one on the thigh and one on the back) for 7 days at home, at baseline, after 8-14 weeks (according to the muncipality) and after 52 weeks.

SECONDARY OUTCOMES:
Changes in VO2-peak from baseline to 52 weeks, measured by the standardised walking test (in the InterWalk) | 52 weeks
  VO2-peak is measured by the standardised walking test (in the InterWalk)
Change in Endurance in the lower extremities from baseline to 52 weeks, measured by sit-to-stand (30 seconds) | January 2015 to July 2017
  Endurance in the lower extremities is measured by sit-to-stand (30 seconds)
Changes in Self-rated physical activity from baseline to 52 weeks, measured by "The Resent Physical Activity Questionnaire" (RPAQ) | 52 weeks
  Self-rated physical activity by "The Resent Physical Activity Questionnaire" (RPAQ)
Changes in Health related quality of life from baseline to 52 weeks, measured by SF-12 | 52 weeks
  Health related quality of life by SF-12
Changes in Motivation for physical activity and behaviour change from baseline to 52 weeks, measured by the Behavioural exercise regulation questionnaire (BREQ-2). | 52 weeks
  Motivation for physical activity and behaviour change will be measure by the Behavioural exercise regulation questionnaire (BREQ-2).
Body temperature, measured by an ear thermometer | 52 weeks
  Body temperature will be measured by an ear thermometer, to detect possible mitochondrial effects of exercise.

OTHER OUTCOMES:
Exploratory secondary outcome - Personality (measured once at baseline), measured by the NEO-Five Factor Inventory (NEO-FFI) and a Sensation Seeking Scale (SES). | 12 weeks
  The patient will be asked to complete two questionnaire regarding personality, the NEO-Five Factor Inventory (NEO-FFI) and a Sensation Seeking Scale (SES).
  We do not know much about what characterizes the individual to either participate or to decline an intervention e.g. diet, smoking cessation or physical activity. The two personality questionnaires are part of the project because it is essential to get more knowledge on personality traits, risk behavior and adherence to an intervention in this case physical activity. By this knowledge it will be possible to better individualize the intervention and by this hopefully get a higher adherence in the long term.
Changes in physical activity habits and diabetic motivation from baseline to 52 weeks - patients will be asked to answer 4 questions regarding their physical activity habits | 52 weeks
  Changing habits is difficult and when having a lifestyle disease it can be even more difficult. It is important to get knowledge on the diabetic motivation for the physical activity habits when being diagnosed with type 2 diabetes.
  The patients will be asked to answer 4 questions regarding their physical activity habits at baseline, after 8-14 weeks (according to the municipality) and after 52 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Laura S Valentiner, Principal Investigator — University of Copenhagen
Locations (1):
- University of Copenhagen, Copenhagen, Denmark

REFERENCES:
- [Background] Shaw JE, Sicree RA, Zimmet PZ. Global estimates of the prevalence of diabetes for 2010 and 2030. Diabetes Res Clin Pract. 2010 Jan;87(1):4-14. doi: 10.1016/j.diabres.2009.10.007. Epub 2009 Nov 6. PMID 19896746
- [Background] Unwin N, Gan D, Whiting D. The IDF Diabetes Atlas: providing evidence, raising awareness and promoting action. Diabetes Res Clin Pract. 2010 Jan;87(1):2-3. doi: 10.1016/j.diabres.2009.11.006. Epub 2009 Dec 4. No abstract available. PMID 19962207
- [Background] Sorensen HT, Friborg S, Rungby J, Christensen JS, Vaag A, Beck-Nielsen H. The Danish national type 2 diabetes cohort - the DD2 study. Clin Epidemiol. 2012;4(Suppl 1):1-5. doi: 10.2147/CLEP.S31104. Epub 2012 Sep 21. No abstract available. PMID 23152706
- [Background] Pal K, Eastwood SV, Michie S, Farmer AJ, Barnard ML, Peacock R, Wood B, Inniss JD, Murray E. Computer-based diabetes self-management interventions for adults with type 2 diabetes mellitus. Cochrane Database Syst Rev. 2013 Mar 28;2013(3):CD008776. doi: 10.1002/14651858.CD008776.pub2. PMID 23543567
- [Background] Thomsen RW, Friborg S, Nielsen JS, Schroll H, Johnsen SP. The Danish Centre for Strategic Research in Type 2 Diabetes (DD2): organization of diabetes care in Denmark and supplementary data sources for data collection among DD2 study participants. Clin Epidemiol. 2012;4(Suppl 1):15-9. doi: 10.2147/CLEP.S30082. Epub 2012 Sep 21. PMID 23071407
- [Background] Pouwer F, Geelhoed-Duijvestijn PH, Tack CJ, Bazelmans E, Beekman AJ, Heine RJ, Snoek FJ. Prevalence of comorbid depression is high in out-patients with Type 1 or Type 2 diabetes mellitus. Results from three out-patient clinics in the Netherlands. Diabet Med. 2010 Feb;27(2):217-24. doi: 10.1111/j.1464-5491.2009.02903.x. PMID 20546267
- [Background] Lloyd CE, Hermanns N, Nouwen A, Pouwer F, Underwood L, Winkley K. The epidemiology of depression and diabetes: In: Katon W, May M, Sartorius N, eds. Depression and Diabetes.Oxford:Wiley-Blackwell, 2010
- [Background] Boule NG, Haddad E, Kenny GP, Wells GA, Sigal RJ. Effects of exercise on glycemic control and body mass in type 2 diabetes mellitus: a meta-analysis of controlled clinical trials. JAMA. 2001 Sep 12;286(10):1218-27. doi: 10.1001/jama.286.10.1218. PMID 11559268
- [Background] Karstoft K, Winding K, Knudsen SH, Nielsen JS, Thomsen C, Pedersen BK, Solomon TP. The effects of free-living interval-walking training on glycemic control, body composition, and physical fitness in type 2 diabetic patients: a randomized, controlled trial. Diabetes Care. 2013 Feb;36(2):228-36. doi: 10.2337/dc12-0658. Epub 2012 Sep 21. PMID 23002086
- [Background] Di Loreto C, Fanelli C, Lucidi P, Murdolo G, De Cicco A, Parlanti N, Ranchelli A, Fatone C, Taglioni C, Santeusanio F, De Feo P. Make your diabetic patients walk: long-term impact of different amounts of physical activity on type 2 diabetes. Diabetes Care. 2005 Jun;28(6):1295-302. doi: 10.2337/diacare.28.6.1295. PMID 15920042
- [Background] Sone H, Tanaka S, Iimuro S, Tanaka S, Oida K, Yamasaki Y, Oikawa S, Ishibashi S, Katayama S, Yamashita H, Ito H, Yoshimura Y, Ohashi Y, Akanuma Y, Yamada N; Japan Diabetes Complications Study Group. Long-term lifestyle intervention lowers the incidence of stroke in Japanese patients with type 2 diabetes: a nationwide multicentre randomised controlled trial (the Japan Diabetes Complications Study). Diabetologia. 2010 Mar;53(3):419-28. doi: 10.1007/s00125-009-1622-2. Epub 2010 Jan 7. PMID 20054522
- [Background] Pedersen BK, Saltin B. Evidence for prescribing exercise as therapy in chronic disease. Scand J Med Sci Sports. 2006 Feb;16 Suppl 1:3-63. doi: 10.1111/j.1600-0838.2006.00520.x. PMID 16451303
- [Background] Avery L, Flynn D, van Wersch A, Sniehotta FF, Trenell MI. Changing physical activity behavior in type 2 diabetes: a systematic review and meta-analysis of behavioral interventions. Diabetes Care. 2012 Dec;35(12):2681-9. doi: 10.2337/dc11-2452. PMID 23173137
- [Background] Plotnikoff RC, Costigan SA, Karunamuni ND, Lubans DR. Community-based physical activity interventions for treatment of type 2 diabetes: a systematic review with meta-analysis. Front Endocrinol (Lausanne). 2013 Jan 29;4:3. doi: 10.3389/fendo.2013.00003. eCollection 2013. PMID 23372566
- [Background] Conn VS, Hafdahl AR, Mehr DR, LeMaster JW, Brown SA, Nielsen PJ. Metabolic effects of interventions to increase exercise in adults with type 2 diabetes. Diabetologia. 2007 May;50(5):913-21. doi: 10.1007/s00125-007-0625-0. Epub 2007 Mar 7. PMID 17342472
- [Background] Barnard KD, Peyrot M, Holt RI. Psychosocial support for people with diabetes: past, present and future. Diabet Med. 2012 Nov;29(11):1358-60. doi: 10.1111/j.1464-5491.2012.03727.x. No abstract available. PMID 22681530
- [Background] Beck-Nielsen H, Henriksen JE. [Type 2 diabetes in Denmark]. Ugeskr Laeger. 2012 Sep 10;174(37):2132-8. Danish. PMID 22971291
- [Background] de Jongh T, Gurol-Urganci I, Vodopivec-Jamsek V, Car J, Atun R. Mobile phone messaging for facilitating self-management of long-term illnesses. Cochrane Database Syst Rev. 2012 Dec 12;12(12):CD007459. doi: 10.1002/14651858.CD007459.pub2. PMID 23235644
- [Background] Colberg SR, Sigal RJ, Fernhall B, Regensteiner JG, Blissmer BJ, Rubin RR, Chasan-Taber L, Albright AL, Braun B; American College of Sports Medicine; American Diabetes Association. Exercise and type 2 diabetes: the American College of Sports Medicine and the American Diabetes Association: joint position statement executive summary. Diabetes Care. 2010 Dec;33(12):2692-6. doi: 10.2337/dc10-1548. No abstract available. PMID 21115771
- [Background] Little JP, Jung ME, Wright AE, Wright W, Manders RJ. Effects of high-intensity interval exercise versus continuous moderate-intensity exercise on postprandial glycemic control assessed by continuous glucose monitoring in obese adults. Appl Physiol Nutr Metab. 2014 Jul;39(7):835-41. doi: 10.1139/apnm-2013-0512. Epub 2014 Feb 18. PMID 24773254
- [Background] El-Gayar O, Timsina P, Nawar N, Eid W. Mobile applications for diabetes self-management: status and potential. J Diabetes Sci Technol. 2013 Jan 1;7(1):247-62. doi: 10.1177/193229681300700130. PMID 23439183
- [Background] El-Gayar O, Timsina P, Nawar N, Eid W. A systematic review of IT for diabetes self-management: are we there yet? Int J Med Inform. 2013 Aug;82(8):637-52. doi: 10.1016/j.ijmedinf.2013.05.006. Epub 2013 Jun 21. PMID 23792137
- [Background] Ahlin K, Billhult A. Lifestyle changes - a continuous, inner struggle for women with type 2 diabetes: a qualitative study. Scand J Prim Health Care. 2012 Mar;30(1):41-7. doi: 10.3109/02813432.2011.654193. Epub 2012 Feb 12. PMID 22324486
- [Background] Malpass A, Andrews R, Turner KM. Patients with Type 2 Diabetes experiences of making multiple lifestyle changes: a qualitative study. Patient Educ Couns. 2009 Feb;74(2):258-63. doi: 10.1016/j.pec.2008.08.018. Epub 2008 Oct 9. PMID 18848413
- [Background] Welschen LM, van Oppen P, Dekker JM, Bouter LM, Stalman WA, Nijpels G. The effectiveness of adding cognitive behavioural therapy aimed at changing lifestyle to managed diabetes care for patients with type 2 diabetes: design of a randomised controlled trial. BMC Public Health. 2007 May 8;7:74. doi: 10.1186/1471-2458-7-74. PMID 17488511
- [Background] Sarkar U, Fisher L, Schillinger D. Is self-efficacy associated with diabetes self-management across race/ethnicity and health literacy? Diabetes Care. 2006 Apr;29(4):823-9. doi: 10.2337/diacare.29.04.06.dc05-1615. PMID 16567822
- [Background] Centis E, Trento M, Dei Cas A, Pontiroli AE, De Feo P, Bruno A, Sasdelli AS, Arturi F, Strollo F, Vigili De' Kreutzenberg S, Invitti C, Di Bonito P, Di Mauro M, Pugliese G, Molteni A, Marchesini G. Stage of change and motivation to healthy diet and habitual physical activity in type 2 diabetes. Acta Diabetol. 2014 Aug;51(4):559-66. doi: 10.1007/s00592-013-0551-1. Epub 2014 Jan 20. PMID 24442514
- [Background] Ekelund U, Brage S, Griffin SJ, Wareham NJ; ProActive UK Research Group. Objectively measured moderate- and vigorous-intensity physical activity but not sedentary time predicts insulin resistance in high-risk individuals. Diabetes Care. 2009 Jun;32(6):1081-6. doi: 10.2337/dc08-1895. Epub 2009 Feb 27. PMID 19252168
- [Background] Beck-Nielsen H, Solomon TP, Lauridsen J, Karstoft K, Pedersen BK, Johnsen SP, Nielsen JS, Kryger TB, Sortso C, Vaag A. The Danish Centre for Strategic Research in Type 2 Diabetes (DD2) study: expected outcome from the DD2 project and two intervention studies. Clin Epidemiol. 2012;4(Suppl 1):21-6. doi: 10.2147/CLEP.S30655. Epub 2012 Sep 21. PMID 23071408
- [Background] Jones CJ, Rikli RE, Beam WC. A 30-s chair-stand test as a measure of lower body strength in community-residing older adults. Res Q Exerc Sport. 1999 Jun;70(2):113-9. doi: 10.1080/02701367.1999.10608028. PMID 10380242
- [Background] Besson H, Brage S, Jakes RW, Ekelund U, Wareham NJ. Estimating physical activity energy expenditure, sedentary time, and physical activity intensity by self-report in adults. Am J Clin Nutr. 2010 Jan;91(1):106-14. doi: 10.3945/ajcn.2009.28432. Epub 2009 Nov 4. PMID 19889820
- [Background] Ware J Jr, Kosinski M, Keller SD. A 12-Item Short-Form Health Survey: construction of scales and preliminary tests of reliability and validity. Med Care. 1996 Mar;34(3):220-33. doi: 10.1097/00005650-199603000-00003. PMID 8628042
- [Background] Golubic R, May AM, Benjaminsen Borch K, Overvad K, Charles MA, Diaz MJ, Amiano P, Palli D, Valanou E, Vigl M, Franks PW, Wareham N, Ekelund U, Brage S. Validity of electronically administered Recent Physical Activity Questionnaire (RPAQ) in ten European countries. PLoS One. 2014 Mar 25;9(3):e92829. doi: 10.1371/journal.pone.0092829. eCollection 2014. PMID 24667343
- [Background] Mortensen EL, Flensborg-Madsen T, Molbo D, Christensen U, Osler M, Avlund K, Lund R. Personality in late midlife: associations with demographic factors and cognitive ability. J Aging Health. 2014 Feb;26(1):21-36. doi: 10.1177/0898264313519317. PMID 24584258
- [Background] KOLIN EA, PRICE L, ZOOB I. DEVELOPMENT OF A SENSATION-SEEKING SCALE. J Consult Psychol. 1964 Dec;28:477-82. doi: 10.1037/h0040995. No abstract available. PMID 14242306
- [Background] Schulz KF, Altman DG, Moher D; CONSORT Group. CONSORT 2010 statement: updated guidelines for reporting parallel group randomised trials. BMJ. 2010 Mar 23;340:c332. doi: 10.1136/bmj.c332. PMID 20332509
- [Background] Siegert RJ, Taylor WJ. Theoretical aspects of goal-setting and motivation in rehabilitation. Disabil Rehabil. 2004 Jan 7;26(1):1-8. doi: 10.1080/09638280410001644932. PMID 14660192
- [Background] Meyer PJ. "What would you do if you knew you couldn't fail? Creating S.M.A.R.T. Goals". Attitude is everything: If you want to succeed above and beyond. Meyer Resource Group Incorporated, ISBN 978-0-89811-304-4
- [Derived] Thorsen IK, Yang Y, Valentiner LS, Glumer C, Karstoft K, Brond JC, Nielsen RO, Brons C, Christensen R, Nielsen JS, Vaag AA, Pedersen BK, Langberg H, Ried-Larsen M. The Effects of a Lifestyle Intervention Supported by the InterWalk Smartphone App on Increasing Physical Activity Among Persons With Type 2 Diabetes: Parallel-Group, Randomized Trial. JMIR Mhealth Uhealth. 2022 Sep 28;10(9):e30602. doi: 10.2196/30602. PMID 36170002
- [Derived] Valentiner LS, Ried-Larsen M, Karstoft K, Brinklov CF, Brons C, Nielsen RO, Christensen R, Nielsen JS, Vaag AA, Pedersen BK, Langberg H. Long-term effect of smartphone-delivered Interval Walking Training on physical activity in patients with type 2 diabetes: protocol for a parallel group single-blinded randomised controlled trial. BMJ Open. 2017 Apr 7;7(4):e014036. doi: 10.1136/bmjopen-2016-014036. PMID 28389489